CLINICAL TRIAL: NCT01258621
Title: Learning Curve for Laparoscopic Distal Pancreatectomy in a High-volume Hospital
Brief Title: Learning Curve for Laparoscopic Distal Pancreatectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Università Vita-Salute San Raffaele (Other)
Responsible Party: Marco Braga, MD, Università Vita-Salute San Raffaele
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PANCREAS-LDP2010
Record Dates: First submitted 2010-12-10; First posted 2010-12-13 (Estimated); Last update posted 2010-12-13 (Estimated); Status verified 2010-08

CONDITIONS: Pancreatic Lesions Located at Body or Tail.
Keywords: distal pancreatectomy, laparoscopy, learning curve
MeSH Terms: interventions — Laparoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Laparoscopic Distal Pancreatectomy (Experimental)
  Interventions: Procedure: Laparoscopy

INTERVENTIONS:
Procedure: Laparoscopy — Laparoscopic distal pancreatectomy

SUMMARY:
Laparoscopic distal pancreatectomy (LDP) for benign and borderline pancreatic lesions has recently becoming the treatment of choice in experienced centres. No data have been published about learning curve so far. The purpose of this study was to identify the learning curve period for performing LDP.

DETAILED DESCRIPTION:
Between March 2009 and August 2010 all patients with lesion of body or tail of pancreas were assessed for eligibility for LDP. Exclusion criteria were: major vessels contact in cancer patients, severe organ dysfunction, BMI > 35, and refusing laparoscopic approach. All laparoscopic procedures were carried out by the same surgical team with large experience in open pancreatic surgery. All patients were treated according to an early recovery after surgery protocol. Primary endpoint was conversion rate. Secondary endpoints were operation time, operative blood loss, postoperative morbidity, and length of stay.

ELIGIBILITY:
Inclusion Criteria:

* pancreatic lesion located at body or tail

Exclusion Criteria:

* major vessels infiltration
* severe organ dysfunction
* refusing laparoscopic approach

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-03; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Conversion to open surgery | during surgery; 3 to 5 hours from the start of the procedure

SECONDARY OUTCOMES:
Operative Time | during surgery; 3 to 5 hours from the start of the procedure
Blood loss | during surgery; 3 to 5 hours from the start of the procedure
Length of Hospital Stay | Postoperative. From 0 to 30 days after discharge.

CONTACTS AND LOCATIONS:
Locations (1):
- San Raffaele Hospital, Milan, Italy